CLINICAL TRIAL: NCT04784962
Title: Neuromuscular Stimulation for Rehabilitation After General and Vascular Surgery - a Pilot Randomised Clinical Study
Brief Title: NMES for Rehab After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P84082; 281309 (Other: National Research Ethics Service (IRAS)); 20CX6284 (Other: Institutional JRCO Assessment Number)
Record Dates: First submitted 2021-02-23; First posted 2021-03-05 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Surgery; Vascular Diseases
Keywords: rehabilitation
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sham and active devices are identical and will be randomly allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Sham Comparator): Sham device
  Interventions: Device: Revitive Medic Neuromuscular Stimulation Device (Sham)
- Intervention Arm (Experimental): Standard rehabilitation care including physiotherapy + Adjunctive Neuromuscular Stimulation Device Usage
  Interventions: Device: Revitive Medic Neuromuscular Stimulation Device

INTERVENTIONS:
Device: Revitive Medic Neuromuscular Stimulation Device — Usage of the Revitive NMES device - 1-6 sessions daily (30 minutes per session).
  Arms: Intervention Arm
Device: Revitive Medic Neuromuscular Stimulation Device (Sham) — Usage of the Sham Revitive NMES device - 1-6 sessions daily (30 minutes per session)
  Arms: Control Arm

SUMMARY:
A randomised pilot study assessing the acceptability and feasibility of utilising neuromuscular stimulation devices to enhance post-operative rehabilitation and recovery after general, vascular and urological surgery procedures.

DETAILED DESCRIPTION:
Patients undergoing inpatient rehabilitation after general, vascular or urological surgery will be invited to take part in a randomised study utilising either sham or active neuromuscular stimulation devices to enhance post-operative rehabilitation and physiotherapy.

ELIGIBILITY:
Inclusion Criteria

* Medically stable after index surgery
* Willing and able to participate in study protocol
* All ethnic groups, male or female above the age of 18 years
* Baseline Rockwood Frailty Score of 3 or greater

Exclusion Criteria

* Inability or unwillingness to participate in trial
* Implanted electrical device such as Pacemaker or defibrillator.
* Pregnant
* Acute deep vein thrombosis
* Previous use of NMES device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Safety and Acceptability of NMES as an adjunct for rehabilitation | At discharge from hospital (completion of study) - up to 28 days
  Qualitiative assessment of participant satisfaction and acceptance of NMES device as an adjunct to standard rehabilitation via semi-structured interview

SECONDARY OUTCOMES:
Time to return to baseline mobility and independence | At discharge from hospital (completion of study) - up to 28 days
  Time in days to return to pre-operative mobility and independence
Generic Quality of life - SF-36 | At discharge from hospital (completion of study) - up to 28 days
  Generic quality of life values at entry and exit of study utilising the Short Form 36 health profile
Generic Quality of life - EQ-5D | At discharge from hospital (completion of study) - up to 28 days
  Generic quality of life values at entry and exit of study utilising the EuroQol 5 Domain (EQ-5D) Health Metric
Generic Quality of life - EQ VAS | At discharge from hospital (completion of study) - up to 28 days
  Generic quality of life values at entry and exit of study utilising the EuroQol Visual Analogue Scale
Functional Independence Measure | At discharge from hospital (completion of study) - up to 28 days
  Scoring tool of ability to function independently at entry and exit of study
Barthel Index | At discharge from hospital (completion of study) - up to 28 days
  Scoring tool of independence at entry and exit of study
Rockwood Frailty Index | At discharge from hospital (completion of study) - up to 28 days
  Frailty index scoring tool at entry and exit of study
Satisfaction with device | At discharge from hospital (completion of study) - up to 28 days
  User satisfaction with NMES device assessed by qualitative feedback and assessment
Length of stay | At discharge from hospital (completion of study) - up to 28 days
  Hospital Length of stay
6 Minute Walk | At discharge from hospital (completion of study) - up to 28 days
  Distance walked in 6 minutes at entry and exit of study
Timed Up and Go | At discharge from hospital (completion of study) - up to 28 days
  Time taken to stand and walk from sitting in a chair at entry and exit of study
Compliance with device usage | At discharge from hospital (completion of study) - up to 28 days
  User compliance with NMES device as assessed with usage diary and qualitative feedback
Q Frailty | At discharge from hospital (completion of study) - up to 28 days
  Frailty assessment scale at entry and exit of study
Time taken to achieve - Sitting for >5 minutes | At discharge from hospital (completion of study) - up to 28 days
  Mobility Milestone
Standing for >1 minute | At discharge from hospital (completion of study) - up to 28 days
  Mobility Milestone
Walking >50m | At discharge from hospital (completion of study) - up to 28 days
  Mobility Milestone
Hospital Resource use | At discharge from hospital (completion of study) - up to 28 days
  Contacts with rehabilitation professionals during the using of NMES
Incremental cost-utility ratio, comparing NMES with standard care | At discharge from hospital (completion of study) - up to 28 days
  Cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, DM DSC FRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be available following publication to requesting researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication and analysis complete.
Access Criteria: On request from Academic Institutions

REFERENCES:
- [Derived] Nimura M, Lane T, Rawashdeh M, Onida S, Javed A, Sritharan G, Reese G, Hrouda D, Davies AH. Study protocol for neuromuscular stimulation for rehabilitation after general and vascular surgery: a pilot randomised clinical study. BMJ Open. 2023 Feb 16;13(2):e061800. doi: 10.1136/bmjopen-2022-061800. PMID 36797015